CLINICAL TRIAL: NCT03258060
Title: Cardiac Resynchronisation Therapy In Patients With Narrow QRS Morphology And Heart Failure: Mechanistic Insights From Cardiac MRI And Electroanatomical Mapping
Brief Title: CRT In Narrow QRS Heart Failure: Mechanistic Insights From Cardiac MRI And Electroanatomical Mapping
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: release of other trial indicating futility of this study after recruitment of 1 patient
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: nQRS-CRT
Record Dates: First submitted 2014-03-17; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Pacing; Resynchronization; Electrophysiology; Imaging; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical Dyssynchrony (Active Comparator): Those with cardiac MRI evidence of mechanical dyssynchrony
  Interventions: Procedure: Temporary pacing study; Radiation: Body Surface Mapping
- No Mechanical Dyssynchrony (Active Comparator): Those without mechanical dyssynchrony on cardiac MRI
  Interventions: Procedure: Temporary pacing study; Radiation: Body Surface Mapping

INTERVENTIONS:
Procedure: Temporary pacing study
  Other Names: Electrophysiological study
Radiation: Body Surface Mapping
  Other Names: ECG imaging

SUMMARY:
Cardiac Resynchronisation Therapy (CRT) is a specialist pacemaker procedure that aims to improve the efficiency of the heartbeat. This treatment is used routinely in patients with heart failure and a delay in electrical conduction across the heart seen on the surface ECG (heart tracing). Also CRT has been seen to improve some heart failure patients with a normal electrical conduction (seen on the ECG as a narrow QRS complex). The investigators aim to see if cardiac MRI can be used to select patients with normal electrical conduction for CRT, therefore expanding the number of people who would stand to benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 18 years or above.
  * NYHA grade III-IV heart failure
  * LVEF<35%
  * QRS duration <120ms
  * On optimum medical therapy for heart failure
  * Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
  * Able (in the Investigators opinion) and willing to comply with all study requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* • Female participants who is pregnant, lactating or planning pregnancy during the course of the study.

  * Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
  * Participant who is terminally ill or is inappropriate for placebo medication
  * Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
  * Contraindication to an MRI scan
  * Rate uncontrolled atrial fibrillation precluding a cMR
  * Significant peripheral vascular disease precluding an EP study
  * A contraindication to anticoagulation
  * A prosthetic aortic or tricuspid valve
  * Significant Aortic valve disease
  * Known LV thrombus
  * Insufficient capacity to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04; Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
LV dP/dT during pacing | during temporary pacing study, approximately 2 hours
  To assess LV dP/dT during different pacing modalities by intraventricular pressure wire. A dP/dT change of >10% from baseline is a positive result.

SECONDARY OUTCOMES:
Correlation of electrical and mechanical dyssynchrony | Data is collected prior to temporary pacing study, the post processing needed in order to correlate this data may take up to 2 months
  To correlate the amount of mechanical dyssynchrony seen prior to pacing with electrical dyssynchrony measures from non-contact mapping and body surface mapping

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Rinaldi, MBBS MD FHRS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Department of Cardiovascular Imaging, King's College London, London, United Kingdom